CLINICAL TRIAL: NCT02200029
Title: Open-Label Study With Ademetionine (Heptral®) in Subjects With Intrahepatic Cholestasis (IHC) Associated With Alcoholic Liver Disease (ALD)
Brief Title: Study With Heptral in Subjects With Liver Disease Due to Alcohol Consumption
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: Ascent (Unknown); Datamap (Industry); ClinIntel (Industry); Catalent (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M14-168
Record Dates: First submitted 2014-07-21; First posted 2014-07-25 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Intrahepatic Cholestasis Associated With Alcoholic Liver Disease
Keywords: Intrahepatic Cholestasis
MeSH Terms: conditions — Cholestasis, Intrahepatic | interventions — S-Adenosylmethionine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ademetionine IV (Experimental)
  Interventions: Drug: Ademetionine IV+tablet
- Ademetionine oral (Experimental)
  Interventions: Drug: Ademetionine tablet

INTERVENTIONS:
Drug: Ademetionine IV+tablet — IV ademetionine (500 mg/vial) for 2 weeks followed by oral ademetionine (500 mg/tablet, 2 in the morning and 1 before dinner) for 6 weeks
  Arms: Ademetionine IV
Drug: Ademetionine tablet — oral ademetionine (500 mg/tablet, 2 in the morning and 1 before dinner) for 8 weeks
  Arms: Ademetionine oral

SUMMARY:
A research study of an approved drug called Heptral®, ademetionine, to treat adults with intrahepatic cholestasis (a condition where bile cannot flow from the liver to the duodenum) in pre-cirrhotic and cirrhotic states. Experience from clinical studies in subjects with liver disease has shown that ademetionine is effective.

ELIGIBILITY:
Inclusion criteria:

* Signed informed consent given by the subject
* Age ≥ 18 years to 75 years
* Chronic liver disease due to alcoholic liver disease
* Compensated alcoholic liver disease, defined as having a Maddrey Score < 32 and not being treated with pentoxifylline or prednisolone within 6 months prior to the study
* History of chronic alcohol use, defined as, history of consumption of > 40 g of alcohol per day for females and > 80 g alcohol per day for males for more than 5 years prior to enrolment
* Subjects who abstain from alcohol for more than 2 weeks and will not consume alcohol during the study
* Subjects with Intrahepatic Cholestasis (IHC):
* ALP: more than 1.5 x upper normal limit and
* γGT: more than 3 x upper normal limit
* Subjects with additional serum conjugated bilirubin (SCB) > Upper Limit of Normal (ULN) will be selected for initial IV treatment

Exclusion Criteria:

* Subjects with a known hypersensitivity to the active substance of ademetionine or to any of the inactive ingredients
* Subjects with extrahepatic cause of cholestasis (proven by ultrasound or described in medical history)
* Diagnosis of human immunodeficiency virus (HIV) in medical history
* Subjects with chronic liver disease Child-Pugh class C
* Subjects in the decompensation stage of ALD (such as Maddrey Score >32)
* Subjects with primary sclerosing cholangitis (PSC)
* Subjects with primary biliary cirrhosis (PBC)
* Any form of malignancy within the past 5 years and/or basal cell carcinoma and squamous cell carcinoma of the skin within the past two years
* Subjects with drug-induced liver disease
* History of active substance abuse (oral, inhaled or injected) within one year prior to the study
* Subjects with renal impairment (creatinine level of >2.0 mg/dL or > 150 µmol/l)
* Subjects with known genetic defects affecting the methionine cycle and/or causing homocystinuria and/or hyperhomocysteinemia (e.g., cystathionine beta-synthase deficiency, Vitamin B12 metabolism defect) or known folate, Vitamin B6 or B12 deficiency
* Subjects on total parenteral nutrition in the year prior to screening
* Subjects after or planned for bariatric surgery (jejunoileal bypass or gastric weight loss surgery)
* Subjects after liver transplantation and subjects on the waiting list for liver transplantation
* Subjects with any of the following disease in medical history:
* Viral hepatitis (serum positive HBcAb or Hepatitis C Virus (HCV) RNA)
* Evidence of autoimmune liver disease
* Wilson´s disease
* Hemochromatosis
* Alpha-1-antitrypsin deficiency
* Subjects with history of biliary diversion
* History of major depression or bipolar disease
* Women of childbearing potential: positive urine pregnancy test during screening or unwillingness to use an effective form of birth control during the study.
* Breastfeeding women
* Any condition that, in the opinion of the investigator, does not justify the patient's inclusion into the study
* Investigational drug intake within one month prior to the study
* Active, serious medical disease other than ALD with likely life-expectancy less than five years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Concentrations (Units per liter) of Alkaline phosphatase (ALP) or gamma-glutamyltransferase (γGT) | from baseline up to the end of treatment visit (56-60 days)
  Improvement of ALP or γGT after 8 weeks of treatment with ademetionine compared to baseline

SECONDARY OUTCOMES:
Concentrations of ALP, γGT, Alanine Transaminase (ALT) and Aspartate aminotransferase (AST) (Units per liter) and of serum total and conjugated bilirubin (µmol per liter) | At baseline and after 2 weeks intravenously (IV) treatment or after 4 weeks oral treatment and after 2 months treatment
  Improvement of ALP, γGT and serum total and conjugated bilirubin, ALT and AST compared to baseline
The intensity of clinical symptoms (jaundice, pruritus, fatigue and depressed mood) will be recorded for each symptom separately using six categories: No symptoms (0), minimum (1) to maximum (5). | At baseline and after 2 weeks IV treatment or after 4 weeks oral treatment and after 2 months treatment
  Record of intensity of jaundice, pruritus, fatigue and depressed mood compared to baseline
Evaluation of the responder rate by comparing concentrations at certain time points (units per liter) to baseline concentrations | At baseline and after 2 weeks IV treatment or after 4 weeks oral treatment and after 2 months treatment
  >20% reduction of ALP or γGT or normalization of ALP or γGT compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Suntje Sander-Struckmeier, PhD, Study Director — Abbott
Locations (12):
- Russia (12):
  - Research facility ORG-000962, Moscow
  - Research facility ORG-000957, Moscow
  - Research facility ORG-000961, Moscow
  - Research facility ID ORG-000960, Moscow
  - Research facility ID ORG-000726, Moscow
  - Research facility ORG-000967, Saint Petersburg
  - Research facility ORG-000966, Saint Petersburg
  - Research facility ORG-000968, Saint Petersburg
  - Research facility ORG-000965, Saint Petersburg
  - Research facility ORG-000970, Saint Petersburg
  - Research facility ORG-000958, Troitsk
  - Research facility ORG-000969, Yaroslavl